CLINICAL TRIAL: NCT06833502
Title: Phase II Study of Systemic Screening in Pathologic Node Positive Breast Cancer Following Neoadjuvant Chemotherapy and Surgery
Brief Title: Phase II Study of Systemic Screening in Pathologic Node Positive Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MCC-23433
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Node-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triple negative (Other): Participants diagnosed with triple negative breast cancer.
  Interventions: Other: CT Scan
- HER2+ (Other): Participants diagnosed with HER2+ breast cancer.
  Interventions: Other: CT Scan
- Hormone receptor (HR)+ (Other): Participants diagnosed with hormone receptor (HR)+ breast cancer.
  Interventions: Other: CT Scan

INTERVENTIONS:
Other: CT Scan — Participants will undergo a screening CT thorax, abdomen, pelvis at baseline prior to adjuvant radiation therapy and additional screening CT thorax, abdomen, and pelvis at 6 months if the baseline CT is found to be negative.

SUMMARY:
The purpose of the study is to determine the frequency of systemic metastasis in node positive breast cancer following chemotherapy and surgery. Participants will be asked to spend about 6 months in this study. Participants will undergo a computed tomography (CT) screening of the thorax, abdomen, and pelvis at baseline prior to adjuvant radiation therapy and another CT screening of the thorax, abdomen, and pelvis at 6 months if the baseline CT is found to be negative.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of breast cancer with documentation of ER/PR/HER2 status.
* HR+ will be defined as ER and/or PR ≥ 10%. To be classified as HER2+ disease, overexpression of HER2 by either IHC or in-situ hybridization is necessary as defined by the ASCO / CAP Guidelines27. Triple negative will be classified as ER and PR <10% and HER2-.
* Node positive HER2+ and triple negative breast cancer (ypN+) following receipt of neoadjuvant chemotherapy. HR+/HER2- patients should have ypN2 or ypN3 disease following receipt of neoadjuvant chemotherapy and surgery.
* Patient must have completed a minimum of 8 weeks of standard neoadjuvant chemotherapy consisting of an anthracycline and/or taxane-based regimen. To include HER2 directed therapy for HER2+ patients.
* Age ≥ 18.
* Life expectancy ≥ 6 months.
* Eastern Cooperative Oncology Group performance status 0 to 2.
* Patients must be able to understand and the willingness to sign an informed consent for study procedures.
* Ability to understand and stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Prior diagnosis of systemic metastases.
* Patients with prior history of non-breast cancer malignancies should have NED ≥ 2 years excluding adequately treated non-melanoma skin cancer, in situ cancer of the cervix or bladder.
* Contraindication towards CT IV contrast.
* Chronic kidney disease stage IV or V or end stage renal disease (CrCl <30 ml/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Systemic Metastasis | Baseline and 6 months
  Proportion of participants with systemic metastasis at baseline and 6 months.

SECONDARY OUTCOMES:
Metastasis Treatment | Up to 12 months
  Number of patients receiving surgery, radiation therapy, and/or systemic therapy to manage metastases.
Metastasis Frequency | Up to 12 months
  Proportion of participants with metastasis up to 12 months from baseline CT.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahmed, Principal Investigator — Moffitt Cancer Center; Matthew Mills, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States